CLINICAL TRIAL: NCT02746380
Title: Multi-center (in Korea and Japan), Double-blind, Randomized, Parallel-group Study to Evaluate the Similarity of Efficacy and Safety of LBAL 40mg Subcutaneous Biweekly Injection to Humira® 40mg Subcutaneous Biweekly Injection, as Adjunctive Therapy to Methotrexate (MTX), in Patients With Active Rheumatoid Arthritis Who Had an Inadequate Response to MTX
Brief Title: A Study Comparing LBAL to Humira® in Subjects With Active Rheumatoid Arthritis Despite Methotrexate Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Collaborators: Mochida Pharmaceutical Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-ALCL002
Record Dates: First submitted 2016-04-05; First posted 2016-04-21 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- LBAL (Experimental): Adalimumab
  Interventions: Drug: LBAL
- Humira® (Active Comparator): Adalimumab
  Interventions: Drug: Humira®

INTERVENTIONS:
Drug: LBAL — Adalimumab
  Arms: LBAL
Drug: Humira® — Adalimumab
  Arms: Humira®

SUMMARY:
This is a randomized, double-blind, parallel group, multicenter clinical study to evaluate the efficacy, safety, pharmacokinetics and immunogenicity of LBAL compared to Humira® in subjects with active Rheumatoid Arthritis despite Methotrexate therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients from 20 years to 75 years of age when signing Informed Consent.
* Diagnosed as having RA (Rheumatoid Arthritis) according to the revised 1987 ACR (American College of Rheumatology) criteria for at least 3 months prior to screening
* Patients who have inadequate response to MTX administered for at least 12 weeks before the beginning of screening period and on a stable dose.

Exclusion Criteria:

* patients with active tuberculosis or latent tuberculosis based on current clinical symptoms, chest X-ray test and IFN-γ release assay at screening
* patients with any of the following concomitant diseases and/or history within 24 weeks before the first administration of investigational products in this study; Serious infectious disease, Opportunistic infection, Chronic or recurrent infectious disease
* patients with any seropositive result for hepatitis B or hepatitis C or HIV
* patients who have any of the following diseases; Sepsis, Demyelinating disorders, Lymphoproliferative disease, Infection with prosthetic joint, Autoimmune diseases other than rheumatoid arthritis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
DAS28-ESR | Week 24
  DAS is a combined index to measure the disease activity in patients with Rheumatoid Arthritis (RA).
  DAS28-ESR is calculated by assessing the number of swollen and tender joints (among 28 joints) and measuring the ESR.

CONTACTS AND LOCATIONS:
Locations (2):
- Mochida Investigational site, Tokyo, Japan
- LGLS Investigational site, Seoul, South Korea